CLINICAL TRIAL: NCT05012722
Title: A Comparison of Arterial Stiffness in Patients With Stable Heart Failure and Stable Chronic Kidney Disease Against Decompensated Heart Failure and Acute Kidney Injury
Brief Title: Arterial Stiffness in Heart Failure and Chronic Kidney Disease
Acronym: ASHFCKD
Status: Completed | Type: Observational
Sponsor: University Hospitals Coventry and Warwickshire NHS Trust (Other)
Responsible Party: Sponsor
Other Study IDs: MJ550021
Record Dates: First submitted 2021-08-02; First posted 2021-08-19 (Actual); Last update posted 2024-06-18 (Actual); Status verified 2024-06

CONDITIONS: Arterial Stiffness
Keywords: Heart Failure; Chronic Kidney Disease
MeSH Terms: conditions — Heart Failure; Renal Insufficiency, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood tests only
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (3):
- Decompensated Heart Failure with reduced ejection fraction (HFrEF): Pulse wave velocity to be measured during hospitalisation phase and repeated 4 weeks after when participant is in a stable state i.e stable (HFrEF)
  Interventions: Diagnostic Test: Sphygmocor CVMS (Atocr Medical, Sydney Australia) PWV measurement
- Decompensated Heart Failure with Preserved ejection fraction (HFpEF): Pulse wave velocity to be measured during hospitalisation phase and repeated 4 weeks after when participant is in a stable state i.e stable (HFpEF)
  Interventions: Diagnostic Test: Sphygmocor CVMS (Atocr Medical, Sydney Australia) PWV measurement
- Acute Kidney Injury in patients with Chronic Kidney Disease stage 3a,3b or 4: Pulse wave velocity to be measured during hospitalisation phase and repeated 4 weeks after when participant is in a stable state i.e. stable Chronic Kidney Disease stage 3a, 3b and 4
  Interventions: Diagnostic Test: Sphygmocor CVMS (Atocr Medical, Sydney Australia) PWV measurement

INTERVENTIONS:
Diagnostic Test: Sphygmocor CVMS (Atocr Medical, Sydney Australia) PWV measurement — All patients included in this study will have a pulse wave velocity measurement measured using SphygmoCor cardiovascular management system (CVMS) (Atocr Medical, Sydney Australia) which is a tonometry-based device used to noninvasively obtain vital cardiovascular data.
  Other Names: No intervention

SUMMARY:
This observational study is assessing the effects that arterial stiffness may have on patients with heart failure (HF) and chronic kidney disease (CKD). Arterial stiffness will be measured by assessing pulse wave velocity (PWV). Carotid- Femoral PWV is the gold standard in measuring arterial stiffness non- invasively. Many studies have shown increasing PWV is a predictor of cardiovascular events, but the significance of increasing PWV as a surrogate marker for the potential worsening (decompensation) of HF or CKD has not been explored.

This study aims to investigate patients with HF and CKD by assessing PWV while in a decompensated state and again when in a stable condition after 4 weeks of discharge to investigate a link between decompensation and rise of arterial stiffness.

The research team aim to recruit 120 patients in this study with 40 patients in each of the 3 groups- heart failure with reduced ejection fraction (HFrEF), heart failure with preserved ejection fraction (HFpEF) and acute kidney injury (AKI). All AKI patients would have had known CKD (stages 3a, 3b or 4).

The study participants will be initially recruited in hospital while admitted in an acute state and tests including bloods, ECG, echocardiography and PWV will be performed. The tests (excluding echocardiography) will be repeated 4 weeks after discharge. There is no intervention in this study.

The study seeks to improve the understanding of the role of the vasculature in the development of acute HF in the two common types- HFrEF and HFpEF. As CKD is a common comorbidity in heart failure patients we felt that a study of the behaviour of arterial stiffness in this cohort will add to this understanding. If arterial stiffness is found to be an important component of the HF syndrome therapeutic interest could be focused at managing arterial stiffness with novel therapy.

DETAILED DESCRIPTION:
Research Objective:

The objective of this study is to identify whether or not patients whom are admitted to hospital with acute decompensated heart failure on a background of stable heart failure or acute kidney injury on a background of stable chronic kidney disease stage 3a,3b or 4 show high pulse wave velocity values when compared to being in a stable condition in the community.

This will help improve the understanding in the pathophysiology of decompensated heart failure and acute kidney injury in CKD.

Scientific Justification:

The role of arterial stiffness in the pathophysiology (in particular, the development) of decompensated heart failure is poorly understood. It is suspected that in some types of heart failure (HFpEF) arterial stiffness may be the driving factor for both acute and chronic types but evidence on this is still incomplete.

CKD is a common comorbidity in heart failure patients- an increase in arterial stiffness in this group with AKI is likely to have an impact on the heart failure in those with both CKD and heart failure.

The study aims to assess whether during the decompensated phases of HF or AKI there is an acute increase in arterial stiffness measured by PWV. If this is indeed found, this study will add to the knowledge on the contribution of arterial resistance to the mechanistic pathophysiology in developing acute HF.

The study is designed to improve the understanding of the contribution of the vasculature to the HF syndrome as well as the contribution of CKD to this. If this study reveals that some types of heart (cardiac) failure are more cardiovascular failure, efforts to develop novel therapies can be then directed at the vascular component too.

It may well reveal also that better risk stratification of heart failure may be possible if vascular stiffness was included within the assessment for heart failure.

Design and Methodology

This is a prospective non-randomised, observational, cohort study.

Patients with decompensated HF or AKI, admitted to cardiac or renal wards at UHCW will be introduced to the study by a member of the research or clinical team once they are deemed to be clinically stable enough to consider this.

Study participants will be screened for eligibility criteria (provided later) and if they meet the inclusion and exclusion criteria they will be approached by a member of the research team to discuss the study, and if interested will be provided a participant information sheet. Written consent will be gained at least 24 hours after the study information is provided If the patient agrees to enrol in the study.

Once the participants are deemed due for discharge within 48 to 72 hours and are clinically stable, a member of the research team will measure their pulse wave velocity using the SphygmoCor CVMS machine (Atcor Medical, Sydney, Australia). Three recordings will be taken for each value and averaged. During their in-patient stay if an up-to date echocardiogram has not been performed in the last 6 months this will be undertaken by a qualified member of staff trained in echocardiography.

Additional tests such as electrocardiograms, baseline blood tests (Full blood count, urea and electrolytes, NT pro BNP and eGFR) and clinical observations (Height, Weight, BMI, Blood Pressure, Oxygen saturations, Heart Rate, Respiratory Rate, Temperature) will be undertaken as part of routine in-patient clinical care- these will be recorded. The time estimated for pulse wave velocity measurements to be taken is estimated at around 15- 20minutes with the patient lying flat on their bed.

Once the participant is discharged they will be asked to attend a follow up visit around 4 weeks after discharge. This could be at either Cardiology Research Suite 4th Floor, UHCW or the City of Coventry Health Centre located at Coventry city-centre. At the follow up visit repeat tests will include routine bloods including NT pro BNP, repeat pulse wave velocity assessment and clinical observations such as blood pressure, heart rate, temperature, height and weight will be recorded. After this follow up visit there will be no further routine follow up of the participant.

Through the hospital CRRS system (medical records) the research team can track if the patient is admitted again with either decompensated heart failure or acute kidney injury and record accurately morbidity or mortality data.

The cohorts of patients will be sub-divided into groups. These groups are decompensated HFrEF, decompensated HFpEF, acute kidney injury in CKD stage 3a,3b or 4, stable HFrEF, stable HFpEF and stable CKD stage 3a, 3b or 4. The patients admitted to hospital will act as their own controls during their follow up visit in a stable condition.

In total the study is looking to recruit 40 participants for each of the 3 groups- decompensated HFrEF, decompensated HFpEF and acute kidney injury on CKD (stage 3a, 3b or 4). In total this means 120 participants during the hospitalisation phase who are then followed up.

During the course of data collection in the study the case report forms will be audited to ensure that the research protocol is being followed. An excel database will be created with patient codes for analysis once data collection is complete.

Inclusion and Exclusion Criteria:

Principal Inclusion Criteria

* Male or Female age ≥60
* Known or documented diagnosis of Heart Failure ( Heart Failure with reduced ejection fraction HFrEF or Heart Failure with preserved ejection fraction HFpEF) on admission or prior to admission. (HFrEF is defined as Left Ventricular ejection fraction (LVEF) of <40%, HFpEF is defined as LVEF >50% as in accordance with the classification by the European Society of Cardiology.)
* Patients on optimal evidence based therapy for heart failure
* Known or documented diagnosis of Chronic Kidney Disease stage 3a, 3b or 4, for minimum period of ≥6 months

Exclusion Criteria

* Severe Peripheral Vascular Disease
* Patients who have had a myocardial infarction or coronary artery bypass surgery within 6 months
* Severe Anaemia Hb 70g/dl
* Dementia or unable to consent lack mental capacity
* Bedbound/ Immobile patients
* Severe Liver Failure
* Severe Chronic Obstructive Pulmonary Disease
* Patients on LTOT (Long Term Oxygen Therapy)
* Renal transplant
* Previous or Current Renal Replacement Therapy (Peritoneal Dialysis or Haemodialysis)
* Sepsis

Ethical issues

This study presents minimal risk to the participants involved. All procedures will have informed patient consent. The assessment of arterial stiffness will be performed using a probe placed on the neck and groin regions which will measure pulse wave velocity (measure of arterial stiffness) by a non-invasive, painless and completely safe process known as tonometry.

Other tests include Electrocardiogram (ECG), transthoracic echocardiography (if not done within 6 months) blood tests all of which pose minimal risk and discomfort (except for minor discomfort during venepuncture for blood tests).

A meeting with patients (Patient & Public Involvement -PPI-meeting) was conducted in December 2020 and valuable feedback was received. The PPI representatives were happy with the current protocol of the study and felt that the tests and timing of the tests did not confer any risk to participants. The lack of intervention would encourage patient participation. PPI feedback was given in the design of the patient information sheet in May 2021.

During the Covid pandemic patients will be asked to return for a second visit to the either the hospital (University Hospital Coventry and Warwickshire (UHCW) Cardiology R&D 4th floor suite) or the Community Heart Failure Clinic on Stoney Staton road, in the Coventry city centre to avoid potential exposure to Covid. Follow up appointments do pose additional strain on existing services. This was discussed at the PPI meeting and the recommendations were that the follow up appointments be kept brief. The research team anticipate that the follow up appointment will last no more than 1 hour. If follow up appointments are missed the research team will rearrange an appointment as soon as possible for the participant.

Legal issues There are no legal issues identified in the study. All of the study methods will be in keeping with good clinical practice NIHR guidance and subjected to standards kept within the Research and Development Department at UHCW.

Management Issues Data collection could be affected by problems with devices such as computers at UHCW or problem with the PWV machine manufactured by SphygmoCor CVMS (Atcor Medical, Sydney, Australia). IT device issues will be rectified by consulting the IT department. For any problems with the Pulse Wave Velocity device, engineering staff at UHCW will be consulted for support.

ELIGIBILITY:
Inclusion Criteria:

Male or Female age ≥60 Known or documented diagnosis of Heart Failure ( Heart Failure with reduced ejection fraction HFrEF or Heart Failure with preserved ejection fraction HFpEF) on admission or prior to admission. HFrEF is defined as Left Ventricular ejection fraction (LVEF) of <40%, HFpEF is defined as LVEF >50% as in accordance with the classification by the European Society of Cardiology.

Patients on optimal evidence based therapy for heart failure Known or documented diagnosis of Chronic Kidney Disease stage 3a, 3b or 4, for minimum period of ≥6 months

-

Exclusion Criteria:

Severe Peripheral Vascular Disease Patients who have had a myocardial infarction or coronary artery bypass surgery within 6 months Severe Anaemia Hb 70g/dl Dementia or unable to consent lack mental capacity Bedbound/ Immobile patients Severe Liver Failure Severe Chronic Obstructive Pulmonary Disease Patients on LTOT (Long Term Oxygen Therapy) Renal transplant Previous or Current Renal Replacement Therapy (Peritoneal Dialysis or Haemodialysis) Sepsis

-

Ages: 60 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants will have either have decompensated heart failure or acute kidney injury in CKD stage 3a,3b or 4 during the hospitalisation phase
Sampling Method: Non-Probability Sample
Enrollment: 119 (Actual)
Dates: Start 2022-01-30 (Actual); Primary Completion 2023-12-13 (Actual); Study Completion 2023-12-13 (Actual)

PRIMARY OUTCOMES:
Pulse Wave Velocity (m/s) | 12 months
  PWV is a measure of arterial stiffness which can be done non invasively at bedside using a device called SphygmoCor CVMS machine (Atcor Medical, Sydney, Australia

SECONDARY OUTCOMES:
Assess the relationship between NYHA heart failure class and PWV | 12 months
  Clinical severity of heart failure with arterial stiffness
Assess the relationship between CKD stage and PWV | 12 months
  Stage of CKD with arterial stiffness
Assess any correlation between non invasive blood pressure & PWV | 12 months
  Brachial cuff blood pressure and its relationship with arterial stiffness

CONTACTS AND LOCATIONS:
Overall Officials: Prithwish Banerjee, MD,FRCP,FESC, Study Chair — Professor of Cardiology and Consultant Cardiologist (Chief Investigator); Mithilesh Joshi, MBChB, Study Director — Cardiology Research Fellow (Sub Investigator)
Locations (1):
- University Hospital Coventry and Warwickshire, Coventry, West Midlands, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided
Data will be audited and monitored by UHCW R&D department

REFERENCES:
- [Derived] Joshi M, Tran P, Barber TM, Khweir L, Appunu K, Ayub W, Banerjee P. Arterial stiffness in acute decompensated heart failure and acute kidney injury: a prospective observational cohort study protocol in a tertiary hospital setting. BMJ Open. 2025 Jun 23;15(6):e097718. doi: 10.1136/bmjopen-2024-097718. PMID 40550719